CLINICAL TRIAL: NCT00371267
Title: Telephone-Delivered Cognitive Behavior Therapy for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F4281-I
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: cognitive behavioral therapy; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Telephone-delivered CBT (Experimental): Telephone-delivered cognitive behavior therapy for pain management
  Interventions: Behavioral: Telephone-delivered Cognitive Behavior Therapy
- Arm 2: Telephone patient education (Active Comparator): Telephone-delivered patient education regarding management of chronic pain
  Interventions: Other: Telephone-delivered Patient Education

INTERVENTIONS:
Behavioral: Telephone-delivered Cognitive Behavior Therapy — Telephone-delivered cognitive behavior therapy for pain management
  Arms: Arm 1: Telephone-delivered CBT
Other: Telephone-delivered Patient Education — Telephone-delivered patient education regarding chronic pain
  Other Names: Patient education regarding pain management
  Arms: Arm 2: Telephone patient education

SUMMARY:
The purpose of this study is to determine whether telephone-delivered cognitive behavior therapy is effective in the treatment of chronic pain. To examine the effectiveness of this approach, a two-arm randomized clinical trial was conducted with 98 individuals, 55 years of age and older, who suffered from chronic pain, recruited from a primary care clinic at the VA Medical Center in San Francisco and affiliated VA Community-based Outpatient Clinics (CBOCs) in Santa Rosa, San Bruno, Ukiah, and Eureka.

DETAILED DESCRIPTION:
Chronic pain represents an epidemic in the United States and a serious public health problem, particularly among adults over the age of 55. In the Veterans Health Administration (VHA), nearly 50% of patients seen in primary care settings report disabling pain symptoms. Persistent pain in older adults is often associated with disability, emotional distress, and increased health care utilization and cost. Since an increase in the number of older adults is anticipated over the next two decades, the problem of chronic pain in this age group will take on increased importance.

Although cognitive behavior therapy (CBT) aimed at improving coping skills is now commonly employed within interdisciplinary pain management programs, access to these interventions is often limited due to the distance from clinical care and disabling impact of pain. In addition, the dropout rate in studies of face-to-face CBT for chronic pain further detracts from its impact in pain management. A telephone-delivered version of CBT for chronic pain overcomes these barriers to access.

To examine the effectiveness of this approach, a two-arm randomized clinical trial was conducted with 98 individuals, 55 years of age and older, who suffered from chronic pain, recruited from a primary care clinic at the VA Medical Center in San Francisco and affiliated VA Community-based Outpatient Clinics (CBOCs) in Santa Rosa, San Bruno, Ukiah, and Eureka. In Study Arm 1, patients received telephone-based cognitive behavior therapy (T-CBT); and in Study Arm 2, patients received pain education (T-ED) matched with Study Arm 1 for amount of contact time. Patients in both groups received 12 sessions of telephone-based individual therapy over a 20-week period. Pain management outcomes were measured at mid-treatment (10 weeks), post-treatment (20 weeks), and at 3-month (32 weeks) and 6-month (46 weeks) follow-up. Outcome variables included measures of pain symptoms, physical limitations, coping, emotional distress, and health-related quality of life. The study hypothesis, assessment methodology, and intervention procedures were based on the cognitive-behavioral model of chronic pain

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must be:

* veterans enrolled in a VA primary care clinic
* at least 55 years of age
* have access to a telephone
* have documented pain for at least the past year
* a pain disorder involving muscle strain and inflammation, trauma to nerves, or central nervous system dysfunction
* Their pain condition must be stable and participants must have no clear indication for specific medical/surgical intervention.

Exclusion Criteria:

Patients were excluded who were:

* psychotic
* cognitively impaired
* show significant suicidal risk (history of multiple suicide attempts or actively suicidal)
* currently abusing alcohol or other drugs, including prescribed opioid pain medications
* voice impairment that would prevent participation in telephone counseling
* visual impairment that would prevent use of the workbook and completion of assessment materials.
* Patients will also be excluded who have an unstable medical condition and clear indication for specific medical/surgical intervention in the near future.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Carmody, PhD, Principal Investigator — VA Medical Center, San Francisco
Locations (1):
- VA Medical Center, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Carmody TP, Duncan CL, Huggins J, Solkowitz SN, Lee SK, Reyes N, Mozgai S, Simon JA. Telephone-delivered cognitive-behavioral therapy for pain management among older military veterans: a randomized trial. Psychol Serv. 2013 Aug;10(3):265-275. doi: 10.1037/a0030944. Epub 2012 Dec 17. PMID 23244028

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Telephone-delivered cognitive behavior therapy for pain management
  Cognitive Behavior Therapy: Telephone-delivered cognitive behavior therapy for pain management
- Arm 2: Telephone-delivered patient education regarding management of chronic pain
  Pain Education: Telephone-delivered education regarding chronic pain
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 48 | 50
Completed | 39 | 32
Not Completed | 9 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 69 (10) | 67.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 47 | 49 | 96
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Short Form-12 Physical Health
Description: Level of physical functioning in daily living, health-related quality of life Range: 0-100; higher score = higher functioning Score: Sum of weighted subscale scores
Time Frame: 46 weeks
Population: Veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Telephone CBT: Telephone-delivered cognitive behavior therapy for pain management
  Cognitive Behavior Therapy: Telephone-delivered cognitive behavior therapy for pain management
- Arm 2: Telephone Patient Education: Telephone-delivered patient education regarding management of chronic pain
  Pain Education: Telephone-delivered education regarding chronic pain
Arm/Group | Arm 1: Telephone CBT | Arm 2: Telephone Patient Education
Number analyzed (Participants) | 48 | 50
units on a scale | 44 (9) | 41 (9)
Statistical Analysis 1: Comparison: Arm 1: Telephone CBT vs Arm 2: Telephone Patient Education; Test type: Superiority or Other; p < 0.27, Mixed Models Analysis

2. Secondary Outcome: Beck Depression Inventory (BDI)-2 Total Score
Description: Measure of symptoms of depression indicating severity of depression Total Score = sum of item scores Range: 0-63; higher scores = greater severity of depression
Time Frame: 46 weeks
Population: Veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Telephone CBT | Arm 2: Telephone Patient Education
Number analyzed (Participants) | 48 | 50
units on a scale | 16 (11) | 17 (10)
Statistical Analysis 1: Comparison: Arm 1: Telephone CBT vs Arm 2: Telephone Patient Education; Test type: Superiority or Other; p < 0.35, Mixed Models Analysis

3. Primary Outcome: Short Form-12 Mental Health
Description: Daily functioning, quality of life Range: 0-100; higher scores = higher level of functioning Score: sum of weighted subscale scores
Time Frame: 46 weeks
Population: Veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Telephone CBT | Arm 2: Telephone Patient Education
Number analyzed (Participants) | 48 | 50
units on a scale | 45 (9) | 46 (10)
Statistical Analysis 1: Comparison: Arm 1: Telephone CBT vs Arm 2: Telephone Patient Education; Test type: Superiority or Other; p < 0.74, Mixed Models Analysis

4. Secondary Outcome: Pain Behavior Checklist Total Score
Description: Assessment of behavioral expression of pain Total Score = mean of item scores Range: 0-6; higher = more pain behavior
Time Frame: 46 weeks
Population: Veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Telephone CBT | Arm 2: Telephone Patient Education
Number analyzed (Participants) | 48 | 50
units on a scale | 2.3 (1.3) | 2.4 (1.3)
Statistical Analysis 1: Comparison: Arm 1: Telephone CBT vs Arm 2: Telephone Patient Education; Test type: Superiority or Other; p = 0.39, Mixed Models Analysis

5. Secondary Outcome: Pain Intensity Rating
Description: Measure of rated pain intensity Score = mean Range: 0-5; higher scores = more intense pain
Time Frame: 46 weeks
Population: Veterans with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Telephone CBT | Arm 2: Telephone Patient Education
Number analyzed (Participants) | 48 | 50
units on a scale | 3.6 (1.3) | 3.4 (1.3)
Statistical Analysis 1: Comparison: Arm 1: Telephone CBT vs Arm 2: Telephone Patient Education; Test type: Superiority or Other; p = 0.67, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 46 weeks
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

LIMITATIONS AND CAVEATS:
The fact that the study was conducted in California may have posed some threat to external validity when applying these findings to the nationwide VA system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes